CLINICAL TRIAL: NCT06861855
Title: Prognostic Impact of Immunohistochemical Expression of METTL-14 in Endometrial Carcinoma
Brief Title: Prognosis of METTL-14 in Endometrial Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Ashraf Alfy, Principal investigator, Assiut University
Other Study IDs: prognosisendometrialcarcinoma
Record Dates: First submitted 2025-02-22; First posted 2025-03-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer; Endometrial Adenocarcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endometrial carcinoma
  Interventions: Other: Observation; Behavioral: IHC

INTERVENTIONS:
Other: Observation — observation of METTL-14 prognosis
Behavioral: IHC — IHC of METTL-14

SUMMARY:
1. To evaluate immunohistochemical expression of METTL14 in type1 endometrial carcinoma.
2. To evaluate the correlation between METTL14 expression and clinicopathological parameters of patients with type 1endometrial carcinoma such as tumor grade, lymhovascular invasion, age of pateints, tumor stage, presence of myometrial invasion and presence of cervical stroma affection.
3. To assess correlation of METTL-14 expression with disease free survival and overall survival.

DETAILED DESCRIPTION:
Endometrial cancer(EC) is the second most common gynecologic cancer worldwide(1). In Egypt its incidence rate has increased in recent years, reaching 4.1 per 100,000 women(2). The most common histological subtype is endometrioid adenocarcinoma(3). Endometrial carcinoma can be divided into:Type I and Type II tumors. The incidence of Type I is 60-80% and that of Type II is 20%(4).

N6-methyladenosine (m6A)is the most abundant RNA modification in mammalian mRNA and has a crucial role in the occurrence and development of various diseases, particularly malignant tumors(3). Many factors were found to affect the prognosis of endometrial carcinoma, one of these factors is m6A RNA methylation(5). This modification is dynamic and reversible, and it is catalyzed by three main types of regulators(3). It has been reported that m6A methylation was performed via methyltransferase complex regulators composed of "writer," "eraser," and "reader"(6).

Methyltransferase like 14 (METTL14), a member of "writer", acts to regulate the occurrence of various cancers(7). In most tumors METTL14 acts as an antioncogene, regulating the RNA of genes that help the cell detect and repair DNA damage, acting as a protective mechanism against cancer. Reducing m6A mRNA may be due to METTL14 mutation. Reducing m6A mRNA levels in endometrial cancer cells could enhance cell proliferation and tumorigenicity in vitro and in vivo(8).The role of METTL14 as a risk factor in prognosis of endometrial carcinoma is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Cases of type1endometrial carcinoma with:

  1. Hystrectomy operation
  2. Available full clinical data about patient (age, complaint, findings in clinical examination).
  3. Full data about previous biopsy and radiology.
  4. Full data about patient survival, disease progression and history of chemotherapy for three years.

Exclusion Criteria:

* 1. Any case of type 1 endometrial carcinoma with missing clinical, radiologic or follow up data.

  2. Cases with no available H&E stained slides or formalin fixed paraffin embedded block.

  3.D&C.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: endometrial carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-27 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of immunohistochemical Expression of METTL14 in Type 1 Endometrial Carcinoma | baseline
  Measurement: Percentage of positive METTL14-stained tumor cells using immunohistochemistry (IHC).
  Unit: Percentage (%).
  Time Frame: Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- AssuitU, Asyut, Egypt